CLINICAL TRIAL: NCT06400121
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Single Intravenous Dose, Parallel Efficacy Study of Apimostinel With or Without Subsequent Automated Self-Association Training in Subjects With Major Depressive Disorder
Brief Title: Apimostinel + Automated Neurocognitive Training for Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rebecca Price (Other)
Collaborators: Syndeio Biosciences, Inc (Industry)
Responsible Party: Sponsor-Investigator, Rebecca Price, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY24010064
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Training; Isotonic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Apimostinel + Cognitive Training (Experimental)
  Interventions: Drug: Apimostinel Infusion, Intravenous; Behavioral: Cognitive Training
- Apimostinel + Sham Training (Sham Comparator)
  Interventions: Drug: Apimostinel Infusion, Intravenous; Behavioral: Sham Training
- Placebo + Cognitive Training (Placebo Comparator)
  Interventions: Behavioral: Cognitive Training; Drug: Isotonic Solution, Intravenous

INTERVENTIONS:
Drug: Apimostinel Infusion, Intravenous — Single injection of Apimostinel (10mg)
  Arms: Apimostinel + Cognitive Training; Apimostinel + Sham Training
Behavioral: Cognitive Training — 8 sessions of digital active training
  Arms: Apimostinel + Cognitive Training; Placebo + Cognitive Training
Behavioral: Sham Training — 8 sessions of digital sham training
  Arms: Apimostinel + Sham Training
Drug: Isotonic Solution, Intravenous — Single injection of placebo
  Arms: Placebo + Cognitive Training

SUMMARY:
Apimostinel shows initial promise as a novel rapid-acting antidepressant medication with minimal side effects or safety concerns. Cognitive Training (CT) is a digital intervention that has shown promise in extending the durability of another similar drug (ketamine). This randomized controlled trial will test the efficacy and safety of apimostinel (vs. placebo) for the acute treatment of depression, and will test the potential of CT to enhance and/or extend the durability of apimostinel's antidepressant effect.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of any gender are eligible
2. Aged 18 to 60 years
3. Meets Diagnostic and Statistical Manual, Fifth Edition (DSM-V) criteria for major depressive disorder (MDD)
4. MADRS score ≥ 20 at screening
5. Score >1SD above the normative mean on the Cognitive Triad Inventory (CTI) "self" subscale *OR* <1SD below the normative mean on the Rosenberg self-esteem scale
6. Participants of childbearing potential with a negative serum pregnancy test prior to entry into the study and who are practicing an adequate method of birth control (eg oral or parenteral contraceptives, intrauterine device, barrier, abstinence) and who do not plan to become pregnant during the course of the study. Participants may be included without a negative serum pregnancy test if they are surgically sterile or at least 2 years post- menopausal. Participants who could impregnate a sexual partner should use an acceptable method of birth control during the study, from the day of dosing to 28 days following dose.
7. Participants who could impregnate a partner and their sexual partner of childbearing potential should use an acceptable method of birth control during the study, from day of dosing to 28 days following dose.
8. Clinical laboratory values < 1.5 times the upper limit of normal (ULN) or deemed not clinically significant per the investigator
9. Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments
10. Based on the investigator's clinical judgment, participants with eating disorders, obsessive compulsive disorder (OCD), panic disorder, post-traumatic stress disorder (PTSD), and generalized anxiety disorders secondary to major depressive episodes are permitted.

Exclusion Criteria:

1. Presence of lifetime bipolar, psychotic, or autism spectrum; or current problematic, moderate-to-severe substance use disorder
2. Use of a Monoamine Oxidase Inhibitor (MAOI) within 28 days of infusion date
3. Huntington's, Parkinson's, Alzheimer's, Multiple Sclerosis, or a history of strokes or with one or more seizures without a clear and resolved etiology
4. Currently hospitalized or residing in an in-patient facility during the study participation
5. Acute suicidality or other psychiatric crises requiring treatment escalation, using the Columbia-Suicide Severity Rating Scale (C-SSRS) as both an initial exclusion criteria (C-SSRS "Baseline/Screening" Version for past 1-month period) and as grounds for rescue/removal (C-SSRS "Since Last Visit" form). Participants with C-SSRS suicide ideation scores scored "yes" on items 4 (active suicidal ideation with some intent to act) and/or 5 (active suicidal ideation with specific plan and intent) will be excluded from the study, and if enrolled, will be exited from the study and referred immediately to the nearest emergency mental health facility for additional thorough assessment and appropriate treatment referral.
6. Changes made to treatment regimen within 28 days of drug infusion (Day 0)
7. Reading level <6th grade as per patient self-report
8. Serious, unstable medical illnesses including respiratory [obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics], cardiovascular [including ischemic heart disease and uncontrolled hypertension], and neurologic [including history of severe head injury diagnoses.
9. Clinically significant abnormal findings of laboratory parameters [including urine toxicology screen for drugs of abuse], physical examination, or ECG.
10. Uncontrolled or poorly controlled hypertension, as determined by the study physician's review of vitals collected during screening and any other relevant medical history/records.
11. Patient has clinically significant renal dysfunction as assessed by the estimated glomerular filtration rate <70 mL/min using the Chronic Kidney Disease Epidemiology Collaboration -creatinine methodology.
12. Patient has liver enzyme test results >2 times the upper limit of normal.
13. Patient has resting heart rate (supine) <60 or >100 bpm at the Screening Visit or Pre-Dose Baseline, in the absence of an etiology that, in the judgment of the investigator, is related to exceptionally good cardiovascular fitness.
14. Patient has PR interval >250 msec at the Screening Visit or Pre-Dose Baseline
15. Patients starting hormonal treatment (e.g., estrogen) in the 3 months prior to Screening.
16. Patients taking medications with known activity at the NMDA or AMPA glutamate receptor [e.g., riluzole, amantadine, memantine, topiramate, dextromethorphan (including AuvelityTM), D-cycloserine, ketamine or esketamine], or the mu-opioid receptor.
17. Patients taking any of the following medications: St John's Wort, theophylline, tramadol, metrizamide.
18. Patients who have received ECT in the past 6 months prior to Screening.
19. Patients currently receiving treatment with vagus nerve stimulation (VNS) or repetitive transcranial stimulation (rTMS).
20. Participation in any clinical trial of an investigational product or device within 30 days of enrollment in this trial
21. Positive screen for unreported drugs of abuse, including: cocaine, PCP, opioid or other agent that in the opinion of the investigator is being abused. Positive marijuana screen is not exclusionary if use is consistent with clinical diagnostic interview findings and is seen in the absence of a moderate-to-severe substance use disorder.
22. Participants or sexual partners of participants who are currently pregnant or planning to become pregnant during the course of the study
23. Participants who are breastfeeding
24. History of allergy, sensitivity, or intolerance to apimostinel, zelquistinel, NMDAR ligands including ketamine,dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Trajectories from baseline/screening through 5 days post infusion
  interviewer-rated depression severity, comparing both apimostinel arms (collapsing active and sham CT arms) to placebo+CT arm; range 0-60; high score=worse outcome
Montgomery-Asberg Depression Rating Scale (MADRS) | Trajectories from baseline/screening through 45 days post infusion
  interviewer-rated depression severity, comparing apimostinel+CT to placebo+CT arm; range 0-60; high score=worse outcome

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms | Trajectories from baseline/screening through 45 days post infusion
  Self-reported depression (range: 0-27; higher scores = worse outcome)
Quick Inventory of Depressive Symptoms | Trajectories from baseline/screening through 6 months post infusion
  Self-reported depression (range: 0-27; higher scores = worse outcome)
Montgomery-Asberg Depression Rating Scale (MADRS) | Trajectories from baseline/screening through 6 months post infusion
  interviewer-rated depression severity; range 0-60; high score=worse outcome

OTHER OUTCOMES:
Clinician-Administered Dissociative States Scale (CADSS) | Trajectories from baseline through 120 min post infusion
  Dissociative side effects; range=0-92; higher score=worse outcome
Brief Psychiatric Rating Scale--4 item psychosis subscale (BPRS+) | Trajectories from baseline through 120 min post infusion
  Psychotomimetic side effects; range=4-28; higher score=worse outcome
Time to onset of effect on MADRS | Assessed at each study visit from Day 1 to Month 6
  Defined as the first time the MADRS score is statistically significantly different from placebo group
Duration of effect on MADRS | Assessed at each study visit from Day 1 to Month 6
  Defined as the last time the MADRS score is statistically significantly different from placebo group
Response rate | Assessed at each study visit from Day 1 to Month 6
  Proportion of subjects achieving response (≥ 50% reduction from the baseline MADRS score)
Remission rate | Assessed at each study visit from Day 1 to Month 6
  Proportion of subjects achieving remission (MADRS score ≤ 9)
Maximum decrease in MADRS | Assessed at each study visit from Day 1 to Month 6
  Defined as the mean maximum decrease from baseline in the MADRS at any study timepoint
Time to maximum decrease in MADRS | Assessed at each study visit from Day 1 to Month 6
  Defined as the mean time (in days) at which a participant's maximum decrease from baseline in the MADRS is observed
Columbia Suicide Severity Rating Scale--Suicidal Behavior | Trajectories from baseline/screening through 6 months post infusion
  composite measure of # unique occurrences of any suicidal behavior including: suicide attempts, hospitalization for suicidality, suicide behaviors, or completed suicide
Columbia Suicide Severity Rating Scale--Intensity of Most Severe Ideation | Trajectories from baseline/screening through 6 months post infusion
  suicidal ideation/thoughts; range 0-5; high score=worse outcome
Sedation Scale | Trajectories from baseline through 120 min post infusion
  sedation scale; range 0-4; high score=worse outcome
Implicit Association Test | Trajectories from baseline through 5 days post infusion
  performance-based "target engagement" measure of implicit self-associations; range = -inf-inf; high score=worse outcome
Implicit Association Test | Trajectories from baseline through 45 days post infusion
  performance-based "target engagement" measure of implicit self-associations; range = -inf-inf; high score=worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca B Price, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No